CLINICAL TRIAL: NCT03436251
Title: Evaluation of Local Hyperthermia for the Treatment of Cervical Intraepithelial Neoplasias After 3 Months: a Multicenter, Single-blind, Randomized Controlled Trial
Brief Title: Local Hyperthermia for the Treatment of Cervical Intraepithelial Neoplasias
Acronym: HPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Gao Xinghua, professor, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HH20170606
Record Dates: First submitted 2017-07-22; First posted 2018-02-19 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2020-08

CONDITIONS: Cervical Intraepithelial Neoplasia; Human Papilloma Virus
Keywords: hyperthermia; human papillomavirus virus; cervical intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia; Hyperthermia | interventions — Conization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Local Hyperthermia at 44℃ for HPV+/CIN-1 (Experimental): Local hyperthermia at 44℃ for 30 mins on cervical region, at days of 1,2,3 and 17, 18. HPV+ and normal cytology or HPV+/CIN-1
  Interventions: Device: Local Hyperthermia at 44℃
- local hyperthermia at 37℃ for 30 mins (Sham Comparator): HPV+/CIN-1
  Interventions: Device: Local Hyperthermia at 37℃
- coniztion of the cervix treatment (Active Comparator): coniztion of cervix for HPV+/CIN2, including LEEP or cold knife coniztion
  Interventions: Device: LEEP or cold knife
- Local Hyperthermia at 44℃ for CIN2/HPV+ (Experimental): Local hyperthermia at 44℃ for 30 mins at days of 1,2,3 and 17, 18. HPV+ and CIN2.
  Interventions: Device: Local Hyperthermia at 44℃

INTERVENTIONS:
Device: Local Hyperthermia at 37℃ — As a control, for patients with HPV+/CIN-1 or HPV+ with normal cytology, hyperthermia at 37℃ is applied
  Arms: local hyperthermia at 37℃ for 30 mins
Device: LEEP or cold knife — For patients with HPV+ / CIN-2
  Arms: coniztion of the cervix treatment
Device: Local Hyperthermia at 44℃ — As an experimental arm, for patients with HPV+/CIN-1/CIN2 or HPV+ with normal cytology
  Arms: Local Hyperthermia at 44℃ for CIN2/HPV+; Local Hyperthermia at 44℃ for HPV+/CIN-1

SUMMARY:
Human papillomavirus(HPV) infect epithelial cells and have the capacity to stimulate cell abnormal hyperplasia, especially by those high-risk HPV types. HPV vaccine primarily targeting HPV6/11/16/18 has been available and makes it possible to prevent cervical cancer. However, a large population was left unvaccinated, specifically for those aged ones. In clinic, patients harboring high-risk HPV is quite prevalent in China or other developing nations. Removing the virus and prevention of malignant transformation is required.

Mild local Hyperthermia with a certain temperature range has been successfully used in the treatment of some diseases. It has been utilised in the treatment of some neoplasm, fungal and HPV infections. Investigators' study found that local hyperthermia at 44°C could cleared HPV in more than half of the patients with plantar warts. Investigators also note the fact that in patients with multiple lesions, the clearance of the target lesion is commonly followed by clearance of other distant lesions, a phenomenon suggesting that local hyperthermia could aid in establishing a specific immune response to eliminate HPV.So the purpose of the study is to evaluation local hyperthermia in the treatment of cervical intraepithelial neoplasias grade I and II after 3 months, with positive high-risk type HPVs, and patients with positive testing for high risk HPVs. Appropriate control arms were designed for different conditions.

DETAILED DESCRIPTION:
Mild local Hyperthermia with a certain temperature range has been successfully used in the treatment of some diseases. It has been utilised in the treatment of some neoplasm, fungal and HPV infections. Investigators' study found that local hyperthermia at 44°C could cleared HPV in more than half of the patients with plantar warts. Investigators also note the fact that in patients with multiple lesions, the clearance of the target lesion is commonly followed by clearance of other distant lesions, a phenomenon suggesting that local hyperthermia could aid in establishing a specific immune response to eliminate HPV.So the purpose of the study is to evaluation local hyperthermia in the treatment of cervical intraepithelial neoplasias grade I and II after 3 months, with positive high-risk type HPVs, and patients with positive testing for high risk HPVs. Appropriate control arms were designed for different conditions. One control arm is local hyperthermia at 37°C for 30 mins targeted for CINⅠ, the other control arm is LEEP targeted for CINⅡ. After 3 months, to evaluate the effectivity of local hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old; generally healthy gynecological conditions, normal sexual life; high risk HPV; Cervical biopsy CIN or no cytological changes; signed informed consent

Exclusion Criteria:

* Pregnant woman;local or systematic treatment within 3 months; Comorbidity of other severe gynecological inflammation, infection, or tumor; Comorbidity of other serious illnesses； no guarantee of timely treatment and follow-up

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
clearance rates of HPV | 3 months after the last time of treatment.
  to evaluate the clearance rates in different treatment groups 3 month after treatment.
scoring atypia by cytology/pathology | 3 months after the last time of treatment.
  to evaluate atypia severity score of cervical cells 3 month after treatment.

SECONDARY OUTCOMES:
viral load measurement | 3 months after the last time of treatment.
  to measure the HPV 16 viral load after 3 month of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Gao, Study Director — First Hospital of China Medical University
Locations (1):
- Yang Yang, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Zhang L, Zhang Y, Huo W, Qi R, Guo H, Li X, Wu X, Bai F, Liu K, Qiao Y, Piguet V, Croitoru D, Chen HD, Gao XH. Local Hyperthermia at 44 degrees C Is Effective in Clearing Cervical High-Risk Human Papillomaviruses: A Proof-of-Concept, Randomized Controlled Clinical Trial. Clin Infect Dis. 2021 Nov 2;73(9):1642-1649. doi: 10.1093/cid/ciab369. PMID 33905482